CLINICAL TRIAL: NCT02780297
Title: Prospective Research Rare Kidney Stones (ProRKS)
Acronym: ProRKS
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, PI, Mayo Clinic
Other Study IDs: 16-000494
Record Dates: First submitted 2016-05-11; First posted 2016-05-23 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hyperoxaluria; Cystinuria; Dent Disease; Lowe Syndrome; Adenine Phosphoribosyltransferase Deficiency
Keywords: primary hyperoxaluria; Dent Disease; enteric hyperoxaluria; cystinuria; Lowe Syndrome; Adenine phosphoribosyltransferase deficiency; PH; APRTd; APRT; hyperoxaluria; oxalate; oxalosis; PH type 1; PH type 2; PH type 3; Dents; Dent; Dent 1; Dent 2; APRT deficiency
MeSH Terms: conditions — Hyperoxaluria; Cystinuria; Dent Disease; Oculocerebrorenal Syndrome; Adenine phosphoribosyltransferase deficiency; Hyperoxaluria, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Primary Hyperoxaluria Patients: Patients with confirmed diagnosis of Primary Hyperoxaluria.
- Dent Disease Patients: Patients with confirmed diagnosis of Dent Disease.
- Cystinuria Patients: Patients with confirmed diagnosis of Cystinuria.
- APRT deficiency Patients: Patients with confirmed diagnosis of adenine phosphoribosyltransferase deficiency (APRTd)
- Lowe Syndrome or Dent 2 patients: Patients with confirmed diagnosis of Lowe Syndrome or Dent 2.
- Dent 1 carriers: Patients with confirmed diagnosis of Dent 1. Dent 1 carriers
- Enteric Hyperoxaluria Patients: Patients with confirmed diagnosis enteric hyperoxaluria.

SUMMARY:
The purpose of this study is to determine the natural history of the hereditary forms of nephrolithiasis and chronic kidney disease (CKD), primary hyperoxaluria (PH), cystinuria, Dent disease and adenine phosphoribosyltransferase deficiency (APRTd) and acquired enteric hyperoxaluria (EH). The investigator will measure blood and urinary markers of inflammation and determine relationship to the disease course. Cross-comparisons among the disorders will allow us to better evaluate mechanisms of renal dysfunction in these disorders.

DETAILED DESCRIPTION:
Severe, hereditary forms of nephrolithiasis cause marked excretion of insoluble minerals important in stone formation, including primary hyperoxaluria, cystinuria, Dent disease, and adenine phosphoribosyltransferase deficiency (APRTd). Patients with these disorders experience recurring stones from childhood and are at high risk for chronic kidney disease caused by crystal nephropathy. Enteric hyperoxaluria is an acquired disease characterized by hyperoxaluria and calcium oxalate crystal nephropathy associated with chronic kidney disease, and in that respect similar to the inherited stone diseases. The investigators will collect longitudinal data of individual patients in order to provide clues about potentially modifiable factors that influence disease severity and identify factors leading to kidney injury. the investigator will measure blood and urinary markers of inflammation and determine relationship to the disease course. Cross-comparisons among the disorders will allow to better evaluate mechanisms of renal dysfunction in these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary hyperoxaluria
2. Diagnosis of enteric hyperoxaluria
3. Diagnosis of Dent Disease
4. Diagnosis of Cystinuria
5. Diagnosis of adenine phosphoribosyltransferase deficiency (APRTd)
6. Diagnosis of Lowe Syndrome
7. Diagnosis of Dent Disease Carrier

Exclusion Criteria:

1. Prior renal failure
2. History of liver and/or kidney transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Primary Hyperoxaluria, Dent Disease, Cystinuria and APRT Deficiency, Lowe syndrome, Dent Disease Carriers and Enteric Hyperoxaluria
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
inflammatory blood and urinary biomarkers | Annually for 5 years
  Statistically significant changes (increase or decrease) in inflammatory urinary biomarkers compared to reference values

SECONDARY OUTCOMES:
Longitudinal changes in eGFR | Annually for 5 years
  changes in eGFR during the 5 years

OTHER OUTCOMES:
Development of new onset CKD | Annually for 5 years
  Development of new onset CKD stage 4 (eGFR<30) or stage 5 (eGFR<15)
Lithogenic substances in the urine | Annually for 5 years
  Quantity of change in the substance in the urine
Protein in the urine | Annually for 5 years
  change in protein in the urine
Stone events | Annually for 5 years
  change in number of stone events
Quality of Life | Annually for 5 years
  change in the quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: John Lieske, MD, Principal Investigator — Mayo Clinic
Locations (11):
- United States (8):
  - University of Alabama @ Birmingham, Birmingham, Alabama
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital, Harvard Medical School, Boston, Massachusetts
  - Mayo Clinic Hyperoxaluria Center, Rochester, Minnesota
  - New York University, New York, New York
  - Cincinnati Children's Hosptial Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hosptial of Sick Children, Toronto, Ontario, Canada
- Landspitali Universtiy Hospital, Reykjavik, Iceland
- Shaare Zedek Medica Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials